CLINICAL TRIAL: NCT04294524
Title: Management of Sleep Apnoea Syndrome (SAS) in Patients With Vasovagal Syncope (VVS): a Protocol for the VVS-SAS Registry Study
Brief Title: Management of Sleep Apnoea Syndrome (SAS) in Patients With Vasovagal Syncope (VVS)
Acronym: VVS-SAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PEAS (Pole d'Exploration des Apnees du Sommeil) (Other)
Responsible Party: Principal Investigator, Vincent Puel, Study Director, PEAS (Pole d'Exploration des Apnees du Sommeil)
Other Study IDs: 2017-A03169-44; 2017-A03169-44 (Registry Identifier: RCB number)
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Syncope, Vasovagal; Sleep Apnea Syndromes
MeSH Terms: conditions — Syncope, Vasovagal; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sleep apnea treatment — Sleep apnea treatment as decided according to routine practice. This may be Continuous positive airway pressure (CPAP) or wearing a mandibular advancement device (MAD).

SUMMARY:
This is a multi-centre, registry-based study whose primary objective is to evaluate the effect of treatment for sleep apnoea syndrome (SAS) on the number of syncope/malaise episodes in a population suffering from both idiopathic, recurrent vasovagal syncope/malaises and SAS.

DETAILED DESCRIPTION:
Treatment for sleep apnoea syndrome includes continuous positive airway pressure (CPAP) or a mandibular advancement device (MAD). Additional routine follow-up includes 24 hour holter monitoring on a yearly basis, polysomnography on a yearly basis, multiple sleep latency tests, table tilt tests.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnoea syndrome (>15 respiratory micro awakenings per hour of sleep) with an indication for treatment
* Recurring vasovagal syncope episodes defined as follows: at least three vasovagal syncopes during the last two years - OR- symptoms of orthostatic intolerance occurring in the last 6 months (Symptoms are triggered by orthostatism and can include malaises without loss of consciousness, asthenia, dizziness, visual disturbances, tinnitus, palpitations, headache, limitations of physical activity)

Exclusion Criteria:

* Pathology that may explain syncope symptoms
* Cardiopathy
* Known disautonomia
* Hypotension of known origin
* Adrenal insufficiency
* Thyroid disorder
* History of sudden death in a first degree family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted study population consists of consecutive patients with both vasovagal syncope and sleep apnea syndrome with an indication for treatment.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-02-22 (Estimated); Study Completion 2022-02-22 (Estimated)

PRIMARY OUTCOMES:
Change in 6-month syncope rate | Month -6 to Day 0 versus Months +6 to +12
  Day 0 refers to the initiation of sleep apnea treatment. The baseline syncope rate refers to syncope events occurring between month -6 and day 0 (S_before). The post-treatment syncope rate refers to syncope events occurring between months +6 and +12(S_after). The change is rates is S_before minus S_after.

SECONDARY OUTCOMES:
Syncope/malaise dates | Day 0 to Month 12
  Dates of syncopes/malaises throughout the study.
Patient-reported syncope/malaise frequency | Baseline (Day 0)
  never, rare, every three months, every month, every week, several times per week
Patient-reported syncope/malaise frequency | Yearly visit (month 12)
  never, rare, every three months, every month, every week, several times per week
Patient-reported position of syncopes/malaises | Baseline (Day 0)
  standing, sitting, lying down
Patient-reported position of syncopes/malaises | Yearly visit (month 12)
  standing, sitting, lying down
Patient-reported sycope/malaise trigger | Baseline (Day 0)
  heat, crowding, pain, stress, effort, lack of sleep, none
Patient-reported sycope/malaise trigger | Yearly visit (month 12)
  heat, crowding, pain, stress, effort, lack of sleep, none
Patient-reported sycope/malaise timing | Baseline (Day 0)
  diurnal, nocturnal, postprandial, peri/post-miction/defecation
Patient-reported sycope/malaise timing | Yearly visit (month 12)
  diurnal, nocturnal, postprandial, peri/post-miction/defecation
Patient-reported frequency of signs preceding a loss of consciousness | Baseline (Day 0)
  always, sometimes, never
Patient-reported frequency of signs preceding a loss of consciousness | Yearly visit (month 12)
  always, sometimes, never
VAS for snoring | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for snoring | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nocturnal agitation | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nocturnal agitation | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for restless legs | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for restless legs | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nycturia | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nycturia | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for morning headaches | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for morning headaches | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for absence of libido | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for absence of libido | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nocturnal sweating | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for nocturnal sweating | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for gastro-oesophagien reflux | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for gastro-oesophagien reflux | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for palpitations | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for palpitations | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for lack of concentration while driving | Baseline (Day 0)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
VAS for lack of concentration while driving | Yearly visit (month 12)
  Visual analogue scale (VAS) ranging from 0 (no symptoms) to 10 (strongest symptoms).
12-item Impact of Syncope on Quality of Life (ISQL) questionnaire | Baseline (Day 0)
  The ISQL has a possible range from 0 to 55. Higher scores indicate stronger impact of syncope on quality of life.
12-item Impact of Syncope on Quality of Life (ISQL) questionnaire | Yearly visit (month 12)
  The ISQL has a possible range from 0 to 55. Higher scores indicate stronger impact of syncope on quality of life.
the Epworth Sleepiness Scale | Baseline (Day 0)
  This questionnaire describes sleepiness with a score that ranges from 0 to 24. Higher scores indicate more sleepiness.
the Epworth Sleepiness Scale | Yearly visit (month 12)
  This questionnaire describes sleepiness with a score that ranges from 0 to 24. Higher scores indicate more sleepiness.
Pichot's fatigue scale | Baseline (Day 0)
  This scale describes fatigue and ranges from 0 to 32. Higher scores indicate more fatigue.
Pichot's fatigue scale | Yearly visit (month 12)
  This scale describes fatigue and ranges from 0 to 32. Higher scores indicate more fatigue.
Pichot's depression inventory | Baseline (Day 0)
  This scale ranges from 0 to 13. Higher scores indicate more elements of depression.
Pichot's depression inventory | Yearly visit (month 12)
  This scale ranges from 0 to 13. Higher scores indicate more elements of depression.
Health related quality of life questionnaire (the Medical Outcome Study - Short Form (SF36)) | Baseline (Day 0)
  The SF36 ranges from 0 to 100. Higher scores indicate higher quality of life.
Health related quality of life questionnaire (the Medical Outcome Study - Short Form (SF36)) | Yearly visit (month 12)
  The SF36 ranges from 0 to 100. Higher scores indicate higher quality of life.

OTHER OUTCOMES:
The presence/absence of retrognathia | Baseline (Day 0)
  This is a binary variable indicating qualitative presence or absence of a particular condition.
The presence/absence of archival palate | Baseline (Day 0)
  This is a binary variable indicating qualitative presence or absence of a particular condition.
Mallampati score | Baseline (Day 0)
The presence/absence of anterior open bite | Baseline (Day 0)
  This is a binary variable indicating qualitative presence or absence of a particular condition.
The presence/absence of cervico-mental angle blunting | Baseline (Day 0)
  This is a binary variable indicating qualitative presence or absence of a particular condition.
Body mass index (kg/m2) | Baseline (Day 0)
Abdominal circumference (cm) | Baseline (Day 0)
Systolic blood pressure (mmHg) while lying down | Baseline (Day 0)
Systolic blood pressure (mmHg) while lying down after having remained in a standing position for 3 minutes | Baseline (Day 0)
Diastolic blood pressure (mmHg) while lying down | Baseline (Day 0)
Diastolic blood pressure (mmHg) after having remained in a standing position for 3 minutes | Baseline (Day 0)
Pulse (beats per minute) while lying down | Baseline (Day 0)
Pulse (beats per minute) after having remained in a standing position for 3 minutes | Baseline (Day 0)
Presence/absence of a positive table tilt test | Baseline (Day 0)
  This is a binary variable indicating qualitative presence or absence of a particular condition.
Haemoglobin (g/dl) | Baseline (Day 0)
Haematocrit (%) | Baseline (Day 0)
Blood thyroid stimulating hormone (microU/l) | Baseline (Day 0)
Blood sodium levels (mmol/l) | Baseline (Day 0)
Blood potassium levels (mmol/l) | Baseline (Day 0)
Morning cortisol (mmol/l at 8 am) | Baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Puel, MD, Study Director — Pôle d'exploration des apnées su sommeil (PEAS), Nouvelle Clinique Bel-Air - Bordeaux
Locations (8):
- France (7):
  - University Hospitals of Angers, Angers
  - Clinique Bel Air, Bordeaux
  - University Hospitals of Bordeaux, Bordeaux
  - University Hospitals of Grenoble, Grenoble
  - Clinique Bouchard, Marseille
  - Public Assistance - Hospitals of Marseille, Marseille
  - University Hospitals of Saint Etienne, Saint-Etienne
- Princess Grace Hospital, Monaco, Monaco

REFERENCES:
- [Derived] Puel V, Godard I, Papaioannou G, Gosse P, Pepin JL, Thoin F, Deharo JC, Roche F, Zarqane N, Gagnadoux F, Suehs CM, Molinari N. Management of sleep apnoea syndrome (SAS) in patients with vasovagal syncope (VVS): a protocol for the VVS-SAS cohort study. BMJ Open. 2020 Sep 30;10(9):e038791. doi: 10.1136/bmjopen-2020-038791. PMID 32998925